CLINICAL TRIAL: NCT06476730
Title: Effects of Telerehabilitation Exercise Program on Psychological Health and Delivery Outcomes in Women With Gestational Diabetes Mellitus.
Brief Title: Telerehabilitation Exercise: Effects on Maternal Psychological Health and Delivery Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muzna Haq
Record Dates: First submitted 2024-06-05; First posted 2024-06-26 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Gestational Diabetes; Maternal Psychological Distress
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: There will be two groups, experimental and control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation exercise group (Experimental): This group will receive a structured tele rehabilitation exercise protocol (of low to moderate intensity warm up ,aerobic ,resistance and cool down exercises for 3 times a week progressively increased for 8 weeks) in addition to routine medical care for GDM.
  Interventions: Other: Telerehabilitation exercise program
- Routine medical care (Active Comparator): The control group will receive routine medical care including oral medication, diet and regular walk.
  Interventions: Other: Routine medical care

INTERVENTIONS:
Other: Telerehabilitation exercise program — 5 min warmup will include ankle plantar and dorsiflexion ,trunk side flexion ,shoulder circles ,shoulder ROMS.it will be followed by 5 min aerobics that includes spot marching and side stepping. it will be followed by resistance exercise which will be divided into 3 groups. each group of exercise will be performed one day each. chair squats, arm pulls, seated triceps, biceps curls etc. are included in these resistance exercises. intensity of each exercise will be progressively increased
  Arms: Telerehabilitation exercise group
Other: Routine medical care — The control group will be given routine medical care (including dietary modification, oral anti diabetics (metformin) and advised to do regular walk (20-30min/day).
  Arms: Routine medical care

SUMMARY:
Gestational diabetes occurs when the body can't make enough insulin to manage high blood sugar during pregnancy, usually developing between the 24th and 28th weeks. It affects about 14% of pregnancies worldwide. Women with gestational diabetes often feel more anxious and stressed and have a higher risk of depression during and after pregnancy. This study will explore how telerehabilitation can reduce anxiety and depression and show how exercise can improve the health of pregnant women with gestational diabetes.

DETAILED DESCRIPTION:
The diagnosis of GDM can be unexpected and distressing, leading to feelings of sadness and hopelessness.Women with GDM are at a higher risk of experiencing prenatal and postnatal depression, which can affect their overall well-being and ability to care for their newborn. Regularly checking blood sugar levels, changing diet, and possibly using medication or insulin can be overwhelming. This constant effort and worry about complications can cause a lot of anxiety and stress. Many pregnant women with GDM might not fully understand how exercise can help control their blood sugar levels and improve their overall well-being. Developing a positive attitude towards exercise is important for helping people with gestational diabetes manage their condition effectively through physical activity. The use of telerehabilitation may improve psychological symptoms in participants with GDM.

The control group will receive routine medical care and the experimental group will receive structured telerehabilitation exercise protocol. The results of both groups will be recorded and compared to assess the effectiveness of using telerehabilitation in the treatment of women with GDM in improving psychological health.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 35 years
* Gestational age between 20-28weeks
* diagnosed with Gestational diabetes mellitus through oral glucose tolerance test (OGTT)
* Primigravida and multigravida
* able to do 6 6-minute walk tests under a severity level of 6 on the Borg scale of breathlessness.
* Patients or caregivers have and able to use an electronic device (PC, tablet or smartphone)
* Who signed informed consent

Exclusion Criteria:

* Previously diagnosed T1DM or T2DM
* High-risk pregnancy conditions contraindicating exercise as per ACOG guidelines
* Patients taking insulin regularly.
* Patients with fetal anomalies diagnosed at 20 th week.
* Multiple gestation (twin or triplets).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Center of Epidemiologic studies depression scale (CES-D) | changes from baseline to 8th week
  The CES-DC is an inventory of 20 self-report items regarding depressive symptoms, taking about 5 minutes to completeIn scoring the CES-D, a value of 0, 1, 2 or 3 is assigned to a response depending upon whether the item is worded positively or negatively.Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.
Strait trait anxiety inventory (STAI) | changes from baseline to 8th week
  It is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale.The total score ranges from 0-63.The following guidelines are recommended for the interpretation of scores: 0-9, normal or no anxiety; 10-18, mild to moderate anxiety; 19-29, moderate to severe anxiety; and 30-63, severe anxiety.

SECONDARY OUTCOMES:
Time of delivery | At the time of delivery
  Maternal delivery time in weeks will be noted.
Mode of delivery | At the time of delivery
  Mode of delivery either vaginal or c-section will be noted.
Incidence of instrumental delivery | At the time of delivery
  The incidence of instrumental delivery will be noted wither yes or no.
Incidence of shoulder dystocia | At the time of delivery
  The incidence of shoulder dystocia will be noted wither yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Principal Investigator — Riphah International University, Islamabad, Pakistan
Locations (2):
- Pakistan (2):
  - Pakistan Railways Hospital, Rawalpindi, Punjab Province
  - AlKhidmat Razi Hospital,Rawalpindi, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No